CLINICAL TRIAL: NCT03598751
Title: An International Multicenter Randomized Double-blind Placebo-controlled Clinical Study of the Efficacy and Safety of Subcutaneous BCD-085 in Patients With Psoriatic Arthritis
Brief Title: Clinical Study of Efficacy and Safety of BCD-085 (Monoclonal Anti-IL-17 Antibody) in Psoriatic Arthritis
Acronym: PATERA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCD-085-8
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCD-085 (Experimental): Blinded period:
  BCD-085 120 mg at weeks 0, 1, 2, 4, 6, 8, 10, 14, 18, 22
  Open-label period:
  BCD-085 120 mg at weeks 26, 30, 34, 38, 42, 46, 50, 54
  Interventions: Drug: BCD-085
- Placebo (Placebo Comparator): Blinded period:
  Placebo at weeks 0, 1, 2, 4, 6, 8, 10, 14
  * patients who don't achieve ACR 20 at week 16 will receive BCD-085 at weeks 18 and 22
  * patients who achieve ACR 20 at week 16 will continue placebo at weeks 18 and 22
  Open-label period:
  BCD-085 120 mg at weeks 26, 30, 34, 38, 42, 46, 50, 54
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BCD-085 — 120 mg / 2 mL subcutaneously
  Other Names: Anti-interleukin-17 Monoclonal Antibody
  Arms: BCD-085
Drug: Placebo — 2 mL
  Arms: Placebo

SUMMARY:
Study BCD-085-8/PATERA is a multicentre double-blind placebo-controlled Phase 3 study in patients with psoriatic arthritis (PsA). The objective of the study is to evaluate the efficacy and safety of BCD-085 comparing to placebo in patients with PsA.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent (IC)
* History of psoriatic arthritis (According to CASPAR, 2006) for 6 months
* 3/68 TJC and 3/66 SJC
* RF / ACCP negative
* At least 1 psoriatic plaque ≥ 2 cm and/or psoriatic nails and/or history of confirmed plaque psoriasis
* History of inadequate response to NSAID
* Stable dose of NSAID for 2 weeks
* If on steroids: inadequate response to steroids (at least 3 months of treatment) and stable dose of steroids (10 mg or less) for at least 2 weeks.
* If on MTX: inadequate response to MTX (stable dose 15 - 25 mg / week for at least 2 months)
* In case of history of etanercept therapy: at least 4 weeks after last administration
* In case of history of infliximab therapy: at least 8 weeks after last administration
* In case of history of adalimumab / golimumab / certolizumab pegol therapy: at least 10 weeks after last administration
* In case of history of other mabs / fragments / small molecules : at least 5 half life after last administration
* Negative pregnancy test for women with childbearing potential
* Ability to follow procedures of the study
* Patient and his/her sexual partner with childbearing potential are ready to use reliable contraception, starting at the date of IC sign, within the study period and 4 weeks after the last dose of investigational drug administration. (Not applied to participants/sexual partners who surgically sterilized, and women at menopause for more than 2 years). Reliable contraception considered as 1 barrier method and one of the following: spermicides, oral contraception or intrauterine devices)

Exclusion Criteria:

* Therapy with anti-IL17 / IL17R or anti-IL12/23 or history of therapy with 2 or more monoclonal antibodies or therapy with topical / oral retinoids or phototherapy or other topical medication for psoriasis history or parenteral steroids administration or any intraarticular injections within 4 weeks prior IC sign or any DMARD therapy (excl. methotrexate) on the dated of IC
* Vaccination with live vaccines within 8 weeks prior to IC sign
* Diagnosis of any other chronic infection which may increase the risk of infectious adverse events.
* HIV, HCV, HBV, Syphilis.
* Clinically significant deviations in blood chemistry and blood count
* History of Herpes Zoster
* History of depression, suicidal ideation/behavior.
* Known history of alcohol or drug abuse
* Diagnosis or history of tuberculosis
* Any acute infection or chronic infection flare within 30 days prior to informed consent sign, which may increase (according to the PI opinion) the risk of infectious adverse events.
* Any other documented conditions which increase the risk of AEs development or may interfere with symptoms the disease (masking, increasing or changing) or induce clinical symptoms or laboratory abnormalities similar to PsA:

  1. Uncontrolled diabetes mellitus;
  2. Severe, uncontrolled hypertension;
  3. Presence or history of inflammatory joint disease other than PsA (or any other systemic autoimmune disease (including lupus, Crohn's disease, ulcerative colitis, scleroderma, inflammatory myopathy, mixed connective tissue disease, autoimmune overlap syndrome, fibromyalgia etc.);
  4. History of malignancy, excluding cured basal cell carcinoma / cervical cancer in situ (complete remission for 5 years); cured basal cell skin carcinoma (5 years complete remission), cured ductal breast cancer (5 years complete remission);
  5. Decompensated liver or kidney diseases;
  6. Unstable angina pectoris;
  7. Chronic heart failure, class III-IV according to NYHA;
  8. Myocardial infarction, within 1 year prior to IC sign;
  9. History of organ transplantation;
  10. History of Quincke edema;
  11. History of any significant respiratory diseases, including COPD, asthma or bronchiectasis;
  12. Decompensated respiratory failure;
  13. History of multiple sclerosis,
  14. Devic's disease, or Guillain-Barre syndrome;
  15. Any neurological disease with motor or sensory functions impairment)
* Pregnancy, current or planned in less than 8 weeks after study completion or breastfeeding.
* Simultaneous participation in other clinical trials or participation in other clinical trials with 3 month prior to IC signing date or history of participation it current clinical study (excluding patients dropped out at screening).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
ACR 20 | week 24
  The percentage of patients achieved 20% improvement according to American College of Rheumatology response criteria.
  The ACR Criteria is a dichotomous variable with a positive (=responder) or negative (=non-responder) outcome. The ACR Criteria measures improvement in tender / swollen joint counts and improvement in at least three of the following parameters: 1) patient assessment 2) physician assessment 3) pain scale 4) disability/functional questionnaire 5) acute phase reactant (ESR or CRP). ACR 20 / 50 / 70 has a positive outcome if 20% / 50% / 70% improvement in tender and swollen joint counts was achieved as well as a 20% / 50% / 70% improvement in at least three of the other five criteria.

SECONDARY OUTCOMES:
ACR 20 | Week 1, 2, 4, 8, 12, 16, 20, 24, 30, 38, 46, 54
  The percentage of patients achieved 20% improvement according to American College of Rheumatology response criteria.
ACR 50 | Week 1, 2, 4, 8, 12, 16, 20, 24, 30, 38, 46, 54
  The percentage of patients achieved 50% improvement according to American College of Rheumatology response criteria.
ACR 70 | Week 1, 2, 4, 8, 12, 16, 20, 24, 30, 38, 46, 54
  The percentage of patients achieved 70% improvement according to American College of Rheumatology response criteria.
Proportion of patients achieved PsARC (Psoriatic Arthritis Response Criteria) | Week 1, 2, 4, 8, 12, 16, 20, 24, 30, 38, 46, 54
Change in radiological signs of arthritis (mTSS) | Week 24 and 54
  mTSS - modified Total Sharp Score
Proportion of patients with anti-drug antibodies | Week 2, Week 12, Week 24, Week 38, Week 54

CONTACTS AND LOCATIONS:
Overall Officials: Roman Ivanov, PhD, Study Chair — Biocad
Locations (3):
- 1st City Clinical Hospital, Minsk, Belarus
- Russia (2):
  - Chelyabinsk Regional Clinical hospital, Chelyabinsk
  - North-Western State Medical University n.a. I.I.Mechnikov, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No